CLINICAL TRIAL: NCT00414245
Title: Metformin for the Treatment of Diabetes in Pregnancy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Collaborators: Ben-Gurion University of the Negev (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sor434306ctil
Record Dates: First submitted 2006-12-20; First posted 2006-12-21 (Estimated); Last update posted 2006-12-21 (Estimated); Status verified 2006-12

CONDITIONS: Gestational Diabetes; Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus, Type 2 | interventions — Metformin

INTERVENTIONS:
Drug: metformin

SUMMARY:
The purpose of this study is to determine whether metformin is effective and safe in the treatment of diabetes in pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* GDM A2
* diabetes mellitus type 2
* singleton pregnancy

Exclusion Criteria:

* diabetic nephropathy or proliferative retinopathy
* cannot swallow tablets

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200
Dates: Start 2007-01

PRIMARY OUTCOMES:
glycemic control
pregnancy complications

CONTACTS AND LOCATIONS:
Overall Officials: Boaz Sheizaf, MD, Principal Investigator — division of obstetrics and gynecology, soroka university medical center
Locations (1):
- Division of Obstetrics and Gynecology, Soroka University Medical Center, Beersheba, Israel